CLINICAL TRIAL: NCT01218100
Title: A Randomized, Double-blind, Parallel-Group Study to Evaluate the Effects of First-Line Treatment With a Free Combination of Nebivolol and Lisinopril Compared With Placebo and the Monotherapy Components on Blood Pressure in Patients With Stage 2 Diastolic Hypertension
Brief Title: Efficacy and Safety Study to Evaluate Combination Therapy With Nebivolol and Lisinopril vs. Placebo and Monotherapy in Patients With Stage 2 Diastolic Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEB-MD-25
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Results first posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-05

CONDITIONS: Stage 2 Diastolic Hypertension
MeSH Terms: interventions — Nebivolol; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Combination group - starting dose level nebivolol 5mg and lisinopril 10mg
  Interventions: Drug: nebivolol and lisinopril (free combination)
- 2 (Active Comparator): Nebivolol monotherapy group - starting dose level nebivolol 5mg
  Interventions: Drug: nebivolol monotherapy
- 3 (Active Comparator): Lisinopril monotherapy group - starting dose level lisinopril 10mg
  Interventions: Drug: lisinopril monotherapy
- 4 (Placebo Comparator): Placebo group - starting dose is placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nebivolol and lisinopril (free combination) — nebivolol 5-mg and lisinopril 10-mg (nebivolol non-trade 5-mg tablet and overencapsulated lisinopril 10-mg tablet)/QD/oral administration/up to 12 weeks
  nebivolol 20-mg and lisinopril 40-mg (nebivolol non-trade 20-mg tablet and overencapsulated lisinopril 40-mg tablet)/QD/oral administration/up to 10 weeks
  nebivolol 5-mg and lisinopril 40-mg (nebivolol non-trade 5-mg tablet and overencapsulated lisinopril 40-mg tablet)/QD/oral administration/up to 6 weeks
  nebivolol 20-mg and lisinopril 10-mg (nebivolol non-trade 20-mg tablet and overencapsulated lisinopril 10-mg tablet/QD/oral administration/up to 6 weeks
  Arms: 1
Drug: nebivolol monotherapy — nebivolol 5-mg (non-trade 5-mg tablet)/QD/oral administration/up to 12 weeks
  nebivolol 10-mg (non-trade 10-mg tablet/QD/oral administration/for 1-week down-titration period only)
  nebivolol 20-mg (non-trade 20-mg tablet)/QD/oral administration/up to 10 weeks
  Arms: 2
Drug: lisinopril monotherapy — lisinopril 10-mg (overencapsulated 10-mg tablet)/QD/oral administration/up to 12 weeks lisinopril 40-mg (overencapsulated 40-mg tablet)/QD/oral administration/up to 10 weeks
  Arms: 3
Drug: placebo — Placebo tablet, oral administration/QD/oral administration/up to 12 weeks Placebo capsule, oral administration/QD/oral administration/up to 12 weeks
  Arms: 4

SUMMARY:
This study will evaluate the safety and efficacy of first-line treatment with a free combination (as two separate pills) of nebivolol and lisinopril in patients with stage 2 diastolic hypertension (DBP>= 100 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* male and female outpatients 18 to 64 years of age
* Females must be post-menopausal, or not pregnant and using an approved contraceptive regimen
* stage 2 diastolic hypertension (DBP >= 100 mmHg)

Exclusion Criteria:

* secondary hypertension
* evidence of other concurrent disease or conditions that might interfere with the conduct of the study
* participation in an investigational drug study within 30 days or 5 half-lives, whichever is longer, of Screening (Visit 1).
* have a history of hypersensitivity to nebivolol or other β-blockers, or any contraindication to β-blocker use

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 664 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Stapff, MD PhD, Study Director — Forest Laboratories
Locations (90):
- United States (89):
  - Forest Investigative Site #58, Scottsdale, Arizona
  - Forest Investigative site 080, Tempe, Arizona
  - Forest Investigative site 096, Tucson, Arizona
  - Forest Investigative site 038, Buena Park, California
  - Forest Investigative site 075, Burbank, California
  - Forest Investigative site 042, Costa Mesa, California
  - Forest Investigative site 028, Fountain Valley, California
  - Forest Investigative site 064, Fresno, California
  - Forest Investigative site 079, Lancaster, California
  - Forest Investigative site 097, Long Beach, California
  - Forest Investigative site 049, Los Angeles, California
  - Forest Investigative site 081, Riverside, California
  - Forest Investigative site 040, San Marino, California
  - Forest Investigative site 059, San Ramon, California
  - Forest Investigative site 074, Santa Ana, California
  - Forest Investigative site 072, Tustin, California
  - Forest Investigative site 077, Colorado Springs, Colorado
  - Forest Investigative site 050, Waterbury, Connecticut
  - Forest Investigative site 019, Boca Raton, Florida
  - Forest Investigative site 056, Brandon, Florida
  - Forest Investigative site 043, Brooksville, Florida
  - Forest Investigative site 035, Fort Lauderdale, Florida
  - Forest Investigative site 002, Hialeah, Florida
  - Forest Investigative site 003, Miami, Florida
  - Forest Investigative site 067, Miami, Florida
  - Forest Investigative site 057, Miami, Florida
  - Forest Investigative site 068, Miami, Florida
  - Forest Investigative site 007, Miami, Florida
  - Forest Investigative site 009, New Port Richey, Florida
  - Forest Investigative site 036, Pembroke Pines, Florida
  - Forest Investigative site 005, Pembroke Pines, Florida
  - Forest Investigative site 001, St. Petersburg, Florida
  - Forest Investigative site 004, Tampa, Florida
  - Forest Investigative site 046, Tampa, Florida
  - Forest Investigative site 076, Atlanta, Georgia
  - Forest Investigative site 055, Stockbridge, Georgia
  - Forest Investigative Site 070, Honolulu, Hawaii
  - Forest Investigative site 008, Meridian, Idaho
  - Forest Investigative site 016, Chicago, Illinois
  - Forest Investigative site 085, Chicago, Illinois
  - Forest Investigative site 082, Chicago, Illinois
  - Forest Investigative site 039, Morton, Illinois
  - Forest Investigative site 087, Louisville, Kentucky
  - Forest Investigative site 099, Madisonville, Kentucky
  - Forest Investigative site 060, Owensboro, Kentucky
  - Forest Investigative site 030, New Orleans, Louisiana
  - Forest Investigative site 069, Balitmore, Maryland
  - Forest Investigative site 021, Baltimore, Maryland
  - Forest Investigative site 014, Baltimore, Maryland
  - Forest Investigative site 054, Brockton, Massachusetts
  - Forest Investigative site 095, St Louis, Missouri
  - Forest Investigative site 010, Las Vegas, Nevada
  - Forest Investigative site 012, Las Vegas, Nevada
  - Forest Investigative site 020, Elizabeth, New Jersey
  - Forest Investigative site 065, Asheboro, North Carolina
  - Forest Investigative site 034, Charlotte, North Carolina
  - Forest Investigative site 086, Charlotte, North Carolina
  - Forest Investigative site 089, Hickory, North Carolina
  - Forest Investigative site 094, Hickory, North Carolina
  - Forest Investigative site 027, Lenoir, North Carolina
  - Forest Investigative site 101, Raleigh, North Carolina
  - Forest Investigative site 024, Raleigh, North Carolina
  - Forest Investigative site 013, Shelby, North Carolina
  - Forest Investigative site 022, Winston-Salem, North Carolina
  - Forest Investigative site 098, Cincinnati, Ohio
  - Forest Investigative site 084, Columbus, Ohio
  - Forest Investigative site 026, Dayton, Ohio
  - Forest Investigative site 051, Zanesville, Ohio
  - Forest Investigative site 053, Norman, Oklahoma
  - Forest Investigative site 062, Ashland, Oregon
  - Forest Investigative site 011, Broomall, Pennsylvania
  - Forest Investigative site 061, Philadelphia, Pennsylvania
  - Forest Investigative site 015, Tipton, Pennsylvania
  - Forest Investigative site 045, Cranston, Rhode Island
  - Forest Investigative site 066, Charleston, South Carolina
  - Forest Investigative site 048, Greer, South Carolina
  - Forest Investigative site 093, Mt. Pleasant, South Carolina
  - Forest Investigative site 052, Fayetteville, Tennessee
  - Forest Investigative site 025, Carrollton, Texas
  - Forest Investigative site 006, Houston, Texas
  - Forest Investigative site 029, Houston, Texas
  - Forest Investigative site 047, San Antonio, Texas
  - Forest Investigative site 071, San Antonio, Texas
  - Forest Investigative site 018, Salt Lake City, Utah
  - Forest Investigative site 100, Salt Lake City, Utah
  - Forest Investigative site 023, St. George, Utah
  - Forest Investigative site 031, Norfolk, Virginia
  - Forest Investigative site 041, Norfolk, Virginia
  - Forest Investigative site 078, Tacoma, Washington
- Forest Investigative site 044, Caguas, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 664 patients were randomized to receive double-blind treatment; 661 patients received at least 1 dose of double-blind treatment (Safety Population); and 656 patients had at least 1 postbaseline assessment of trough seated DBP (ITT Population)
Groups:
- Placebo: Placebo group - starting dose is placebo
- Nebivolol + Lisinopril (Combination): Combination group - starting dose level nebivolol 5mg and lisinopril 10mg
- Nebivolol: Nebivolol monotherapy group - starting dose level nebivolol 5mg
- Lisinopril: Lisinopril monotherapy group - starting dose level lisinopril 10mg
Period: Overall Study
Arm/Group | Placebo | Nebivolol + Lisinopril (Combination) | Nebivolol | Lisinopril
Started | 95 | 190 | 189 | 190
Completed | 71 | 165 | 162 | 156
Not Completed | 24 | 25 | 27 | 34
Not completed — Did not meet InclusionExclusion criteria | 1 | 1 | 1 | 2
Not completed — Adverse Event | 4 | 6 | 6 | 7
Not completed — Lack of Efficacy | 9 | 6 | 5 | 12
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 2 | 6 | 7
Not completed — Lost to Follow-up | 3 | 8 | 2 | 1
Not completed — Other Reason | 2 | 2 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nebivolol + Lisinopril (Combination) | Nebivolol | Lisinopril | Total
Number analyzed (Participants) | 95 | 189 | 188 | 189 | 661
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 95 | 189 | 188 | 189 | 661
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.4 (9.7) | 48.8 (8.4) | 49.7 (8.4) | 50.1 (8) | 49.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 75 | 82 | 74 | 278
  Male | 48 | 114 | 106 | 115 | 383
Region of Enrollment [Number; unit: participants]
  United States | 95 | 189 | 188 | 189 | 661

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in Trough Seated Diastolic Blood Pressure at Week 6.
Time Frame: Visit 6/(Week 0) and Visit 9/(Week 6)
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Placebo | Nebivolol + Lisinopril (Combination) | Nebivolol | Lisinopril
Number analyzed (Participants) | 93 | 189 | 185 | 189
mm HG | -8.0 (9.2) | -17.2 (10.2) | -13.3 (8.9) | -12.0 (9.8)

2. Secondary Outcome: The Change From Baseline in Trough Seated Systolic Blood Pressure at Week 6.
Time Frame: Visit 6/(Week 0) and Visit 9/(Week 6)
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Placebo | Nebivolol + Lisinopril (Combination) | Nebivolol | Lisinopril
Number analyzed (Participants) | 93 | 189 | 185 | 189
mm HG | -9.9 (16.4) | -19.2 (19.8) | -14.4 (14.1) | -16.1 (17.2)

ADVERSE EVENTS:
Time Frame: Adverse event reporting occurred from October 6th, 2010 to May 18th, 2011.
Arm/Group | Placebo | Nebivolol + Lisinopril (Combination) | Nebivolol | Lisinopril
Serious Adverse Events (participants affected / at risk) | 2/95 | 2/189 | 3/188 | 4/189
Other Adverse Events (participants affected / at risk) | 15/95 | 31/189 | 32/188 | 24/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=95) | Nebivolol + Lisinopril (Combination) (N=189) | Nebivolol (N=188) | Lisinopril (N=189)
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Vascular disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer perforation (General disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Syncope (Cardiac disorders) | 1 | 0 | 0 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=95) | Nebivolol + Lisinopril (Combination) (N=189) | Nebivolol (N=188) | Lisinopril (N=189)
Upper respiratory tract infection (Infections and infestations) | 4 | 13 | 11 | 8
Nasopharyngitis (Infections and infestations) | 4 | 10 | 12 | 10
Headache (Nervous system disorders) | 8 | 9 | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.